CLINICAL TRIAL: NCT05743075
Title: A Phase III, Randomized, Double-Blind, Placebo-Controlled Clinical Study to Evaluate the Efficacy and Safety of Ensifentrine Over 24 Weeks in Patients With Moderate to Severe Chronic Obstructive Pulmonary Disease
Brief Title: A Study to Evaluate the Efficacy and Safety of Ensifentrine for 24 Weeks in Patients With Moderate to Severe Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Nuance Pharma (shanghai) Co., Ltd (Industry)
Collaborators: Laboratory Corporation of America (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RPL554-CPC001
Record Dates: First submitted 2023-02-14; First posted 2023-02-24 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — ensifentrine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Ensifentrine (Experimental): Eligible subjects will be randomly assigned in a 5:3 ratio to receive either Ensifentrine or placebo. Doses and methods of administration are as follows:
  Ensifentrine (RPL554) 3 mg BID or placebo BID will be administered by aerosol inhalation for 24 weeks; each nebulization time wil be approximately 5 minutes.
  Interventions: Drug: Ensifentrine
- Placebo (Placebo Comparator): Eligible subjects will be randomly assigned in a 5:3 ratio to receive either Ensifentrine or placebo. Doses and methods of administration are as follows:
  Ensifentrine (RPL554) 3 mg BID or placebo BID will be administered by aerosol inhalation for 24 weeks; each nebulization time wil be approximately 5 minutes.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ensifentrine — A dual PDE3/PDE 4 inhibitor
  Arms: Ensifentrine
Drug: Placebo — Placebo solution
  Arms: Placebo

SUMMARY:
This is a multi-center, randomized, double-blind, placebo-controlled, parallel-group clinical study, which aims to evaluate the efficacy, safety, and PK characteristics of Ensifentrine 3 mg twice daily (BID) for 24 weeks treatment of moderate to severe COPD.

DETAILED DESCRIPTION:
The study is divided into 3 periods, a screening/run-in period (run-in for 28 days), a treatment period (24 weeks), and a follow-up period (1 week after the end-of-treatment visit). The qualified subjects will be randomly assigned to the Ensifentrine group or placebo group in a ratio of 5:3, stratified by maintenance therapy in a stable background long-acting muscarinic antagonist (LAMA) or long-acting β2 agonist (LABA) (yes or no) and smoking status (current or past smokers). The Ensifentrine group will receive Ensifentrine 3mg BID nebulizer, and the placebo group will receive placebo nebulizer. The treatment will be lasted given for 24 weeks in both groups.

During treatment, lung function, COPD symptoms, quality of life and other parameters of subjects will be assessed at baseline, week 6, 12, and 24, and the safety will also be assessed over 24-week treatment period and the follow-up period. PK characteristics and dose-response relationship of Ensifentrine will be analyzed for all patients using sparse sampling.

ELIGIBILITY:
Inclusion Criteria:

1. Patient must be 40 to 80 years of age inclusive, at the time of Screening, male or female;
2. Current or former cigarette smokers with a history of cigarette smoking ≥ 10 pack-years;
3. Patients with a clear clinical history of COPD and related symptoms prior to screening;
4. Patients with moderately to severe COPD:

   Pre- and Post- salbutamol FEV1/FVC ratio < 0.70; and Post-salbutamol FEV1 ≥ 30% and ≤ 70% of predicted
5. A score of ≥2 on the Modified Medical Research Council Dyspnea Scale at screening;
6. Patients on no maintenance/background therapy or patients on stable maintenance as either LAMA or LABA therapy.
7. Short-acting β2 agonists (SABAs) should be withheld for at least 6 hours prior to initiation of any spirometry;
8. Female subjects of childbearing potential must have a negative blood pregnancy test 7 days prior to randomization and not be pregnant or lactating. Female subjects of childbearing potential and male subjects with partners of childbearing potential are required to use at least one effective contraceptive method (such as intrauterine contraceptive device, contraceptives or condom) from the screening period, throughout the study period and for at least 30 days after the last dose of blinded investigational product.

Exclusion Criteria:

1. History of life-threatening COPD including Intensive Care Unit admission and/or requiring intubation;
2. Hospitalizations for COPD, pneumonia, or Corona Virus Disease 2019 (COVID-19) in the 12 weeks prior to Screening and/or COPD exacerbation, Newly-occurring pneumonia, a positive COVID-19 test result indicating an active infection before Screening;
3. Patients with lower respiratory tract infection occurred and not resolved within 6 weeks prior to screening and/or prior to randomization;
4. COPD exacerbation requiring oral or parenteral (intravenous, subcutaneous, or intramuscular injection) steroids within 3 months prior to screening;
5. Previous lung resection, OR lung reduction surgery within 1 year of screening;
6. Patients with long term of oxygen use;.
7. Patients with pulmonary rehabilitation;
8. Patients with other respiratory disorders including, but not limited to, current diagnosis of asthma, active tuberculosis, lung cancer, sarcoidosis, pulmonary fibrosis, interstitial lung disease, unstable sleep apnea, known alpha-1 antitrypsin deficiency, cor pulmonale, clinically significant pulmonary hypertension, clinically significant bronchiectasis, or other active pulmonary disease;
9. Major surgery (requiring general anesthesia) within 6 weeks prior to screening;
10. Historical or current evidence of clinically significant cardiovascular disease defined as any disease that in the opinion of the Investigator would put the safety of the patient at risk through participation or which could affect the efficacy or safety analysis if the disease/condition were to exacerbate during the study.
11. Chronic uncontrolled disease including, but not limited to, endocrine, active hyperthyroidism, neurological, hepatic, gastrointestinal, renal, hematological, urological, immunological, psychiatric, or ophthalmic diseases that the investigator believes are clinically significant;
12. Unstable liver disease defined by the presence of ascites, encephalopathy, coagulopathy, hypoalbuminemia, esophageal or gastric varices or persistent jaundice, cirrhosis, known biliary abnormalities (except for Gilbert's syndrome or asymptomatic gallstones);
13. History of malignancy within the past 5 years (except for cured basal cell carcinoma or squamous cell carcinoma of skin, cervical carcinoma in situ), or current potential malignancy under evaluation;
14. Abnormal findings on physical examination that an investigator considers to be clinically significant at screening;
15. Chest X-ray (CXR; posterior-anterior) at screening, or in the 12 months prior to screening with clinically significant abnormalities not attributable to COPD;
16. Electrocardiogram (ECG) finding that is significantly abnormal at Screening;
17. Abnormal lab test result, such as eGFR < 30 mL/min, ALT ≥ 2 × upper limit of normal (ULN), alkaline phosphatase and/or bilirubin > 1.5 × ULN, or any other abnormal hematology, biochemistry, or viral serology deemed by an investigator to be clinically significantly abnormal;
18. Use of an experimental drug within 30 days or 5 half-lives prior to screening (whichever is longer), and/or participation in an interventional clinical trial within 30 days prior to screening;
19. Use of an investigational medical device or participation as a subject in a medical device clinical trial within 30 days prior to screening;
20. Intolerance or hypersensitivity to salbutamol or Ensifentrine (RPL554) or any of its excipients/components;
21. Use of traditional Chinese medicine within 2 weeks prior to first dose of Ensifentrine/ Placebo, which with antispasmodic and anti-asthmatic effects and interfering with respirometry test，that would interfere with the study based on the investigator's discretion;
22. Any other reason that the Investigator considers makes the patient unsuitable to participate.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 526 (Actual)
Dates: Start 2023-03-10 (Actual); Primary Completion 2024-12-06 (Actual); Study Completion 2025-03-07 (Actual)

PRIMARY OUTCOMES:
Average forced expiratory volume in 1 second (FEV1) area under the curve (AUC)0-12h | 12 weeks
  Change from baseline of Average forced expiratory volume in 1 second (FEV1) area under the curve (AUC)0-12h

SECONDARY OUTCOMES:
Peak FEV1 over 4 hours post-dose at Week 12 | 12 weeks
  Change from baseline of Peak FEV1 over 4 hours post-dose at Week 12
Peak FEV1 at Week 6 and Week 24 | 6 or 24 weeks
  Change from baseline peak FEV1
Morning trough FEV1 at Week 6 and Week 24 | 6 or 24 weeks
  Change from baseline morning trough FEV1
Average FEV1 AUC0-4h at Week 6 and Week 24 | 6 or 24 weeks
  Change from baseline average FEV1 AUC0-4h
Average FEV1 AUC0-4h at Week 12 | 12 weeks
  Change from baseline average FEV1 AUC0-4h
Morning trough FEV1 at Week 12 | 12 weeks
  Change from baseline of morning trough FEV1 at Week 12
Evening trough FEV1 at Week 12 | 12 weeks
  Change from baseline of evening trough FEV1 at Week 12
Average FEV1 AUC6-12h at Week 12 | 12 weeks
  Change from baseline of Average FEV1 AUC6-12h at Week 12
Rescue medication use at Weeks 6, 12 and 24 | 6, 12 or 24 weeks
  Change from baseline of Rescue medication use
Evaluating-Respiratory Symptoms (E-RS) Total Score at Weeks 6, 12 and 24 | 6, 12 or 24 weeks
  Change from baseline of Evaluating-Respiratory Symptoms (E-RS) Total Score
SGRQ total score at Weeks 6, 12 and 24 | 6, 12 or 24 weeks
  Change from baseline of SGRQ total score
SGRQ responder analysis at Weeks 6, 12 and 24 | 6, 12 or 24 weeks
  Change from baseline of SGRQ responder analysis
TDI total score at Weeks 6, 12 and 24 | 6, 12 or 24 weeks
  Change from baseline of TDI total score
CAT total score at Weeks 6, 12 and 24 | 6, 12 or 24 weeks
  Change from baseline of CAT total score

CONTACTS AND LOCATIONS:
Locations (1):
- 1st Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No